CLINICAL TRIAL: NCT00261469
Title: Efficacy of Topiramate Prophylaxis as add-on to Triptan Therapy for Migraine
Brief Title: An Open-label Study to Evaluate Topiramate Therapy in Migraine Patients, and Its Effects on Subject Responsiveness to Migraine Treatment With Triptans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005686
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-01

CONDITIONS: Headache
Keywords: Migraine; Headache
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate whether prophylactic use of topiramate (preventative use before a migraine attack) enhances the effectiveness of migraine treatment with triptans.

DETAILED DESCRIPTION:
The objective of this pilot study is to determine if patients with migraine are more responsive to triptans taken for symptomatic headache treatment while on topiramate prophylactic therapy as compared to a baseline period without prophylaxis. The trial is an open-label design, with migraine patients receiving topiramate prophylactically twice a day (maximum of 200 mg/day) for 16 weeks, following a 6-week Prospective Baseline Period.

During the first week of the treatment phase, subjects will begin on a once-daily dose of 25 mg of topiramate at night, and remain on that dose for two weeks. Thereafter, the daily dose will be increased by 25 mg, with twice-daily dosing. If in the investigator's judgement further dosage increases beyond 100 mg/day are indicated, the daily dose will be increased weekly by 25 mg to a daily dose of 150 mg. The daily dose may be increased to a maximum daily dose of 200 mg, if the subject is tolerating the higher doses.

Subjects keep a headache diary in which the following information is recorded: time of onset of headache and indication of type of headache; time headache stops; any symptomatic treatment taken, time that tiptan medication is taken; headache intensity at the time the triptan is taken, 30 minutes, one hour, and two hours post dose; and the presence of nausea at the time the triptan is taken, 30 minutes, on hour, and 2 hours post dose. The primary measure of triptan responsiveness is the proportion of triptan treated migraine attacks that were pain-free at two hours after triptan treatment.

Safety evaluations during the study include the collection of adverse events, laboratory assessments including hematology, chemistry and urinalysis, and vital signs (blood pressure and pulse). The hypothesis is that topiramate prophylaxis will increase the responsiveness of migraine attacks to triptan therapy as measured by the proportion of attacks that are pain-free two hours after triptan therapy. Subjects will begin week 1 of the Topiramate Treatment phase with 25 mg topiramate at night. Thereafter, the dose of topiramate will be increased by 25 mg every second week i.e. week 3 = 50 mg, week 5 =75 mg, week 7 = 100 mg. If, in the investigator's judgment, further dosage increases are indicated, the dose can be increased as follows: week 9 = 125 mg, week 10 = 150 mg, week 11 = 175 mg, week 12 = 200 mgs.The dose may be increased weekly after week 10 if the patient is tolerating the higher.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an established history consistent with migraine, with or without aura, confirming to International Headache Society (HIS) criteria for at least 6 months prior to study entry
* must be using a stable dose of triptan for migraine treatment for at least 3 migraine attacks per month
* must have failed <=2 previous prophylactic medications due to lack of effectiveness
* must have had between 3 and 12 migraine periods and no more than 18 headache days (migraine and non-migraine) during the 6-week Prospective Baseline Period. (A headache day is defined as a calendar day which the subject experienced headache pain for at least 4 hours untreated, or 30 minutes duration treated)
* female subjects who are postmenopausal, surgically incapable of bearing children, or practicing an acceptable method of birth control, and must have a negative pregnancy test at Visit 1.

Exclusion Criteria:

* Subjects with headaches other than migraine with and/or without aura
* onset of migraine after age 50
* overuse analgesics or specific medications for treatment of migraine attacks
* currently on a prophylactic medication for migraine
* history of an unstable medical condition within the past 2 years, malignancy within the past 5 years, major psychiatric disorder within the past 6 months, suicidal ideations or suicide attempt within the past 2 years or history of alcohol or drug abuse within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-04; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The proportion of migraine attacks that are pain-free two hours after triptan treatment, compared to baseline.

SECONDARY OUTCOMES:
Pain relief at two hours after triptan treatment, compared to baseline; the proportion of migraine attacks that are pain-free 1 hour after triptan treatment, compared to baseline; adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- See also: Prophylactic Topiramate and Response to Triptan Treatment for Acute Migraine — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=359&filename=CR005686_CSR.pdf